CLINICAL TRIAL: NCT06137781
Title: Digital Prehabilitation for Patients Undergoing Major Elective Surgery: a Single-arm Pilot Study
Brief Title: Digital Prehabilitation for Patients Undergoing Major Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); PreActiv (Unknown)
Responsible Party: Principal Investigator, Alec Snow, Chief Investigator, Royal United Hospitals Bath NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 333460
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Surgery
Keywords: Prehabilitation; Exercise; Major surgery; Digital health
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Six weeks of digital prehabilitation (Experimental): The digital prehabilitation programme comprises three 35-minute exercise sessions per week, including a warm-up, vigorous intensity aerobic and resistance exercises, and breathing exercises. The digital prehabilitation programme will be tailored to the participant's mobility level and fitness level, which will be assessed via in-platform questionnaires and functional assessments. Functional assessments will be repeated every two weeks to adapt the prehabilitation programme according to changes in fitness level. Within PreActiv's website, participants will be enrolled into a managed community forum of patients and healthcare professionals where they can post their achievements and questions. Alongside access to PreActiv's digital prehabilitation, patients will be given educational materials that summarise the benefits of prehabilitation and how to realise them.
  Interventions: Behavioral: Six weeks of digital prehabilitation

INTERVENTIONS:
Behavioral: Six weeks of digital prehabilitation — All participants will be allocated to receive six weeks of digital prehabilitation via PreActiv's website, plus usual care.

SUMMARY:
Prehabilitation describes the process of improving someone's functional capacity before major surgery. Prehabilitation commonly focuses on exercise training, as fitness level is a predictor of surgical outcomes - the fitter you are before surgery, the lower the risk of complications after surgery. Typically, exercise training is done at the hospital, but research shows that patients would prefer to do prehabilitation exercises in their home.

The goal of this study is to test the feasibility of an online prehabilitation programme made by PreActiv, which can be accessed at home via a website by patients who are awaiting major surgery. PreActiv's prehabilitation programme is six weeks long, and involves three 35-minute exercise sessions per week, with each session including a warm-up, cardio exercises, muscle strengthening exercises, and breathing exercises. Information from this pilot study on the number of exercise sessions attended (adherence) and the number of patients who complete the study (retention) will be used to decide whether we should progress to a larger study that assesses the effectiveness of PreActiv's prehabilitation.

DETAILED DESCRIPTION:
This is a single-arm pilot study to assess the feasibility of PreActiv's digital prehabilitation alongside usual care at the Royal United Hospitals Bath NHS Foundation Trust. The novel provision of tailored, progressive, dynamic, evidence-based, and home-based prehabilitation via PreActiv's digital platform requires evaluation for feasibility, prior to a larger, randomised-controlled trial assessing efficacy. Such research is warranted, as patients indicate a preference to complete prehabilitation at home, rather than at the hospital, but current home-based prehabilitation programmes are one-size-fits-all, and do not adapt to changes in fitness level.

Patients awaiting major surgery and aged 50 years or older will be identified by preoperative nurses and screened by a member of the research team at the Royal United Hospitals Bath NHS Foundation Trust. Eligible patients who provide written informed consent will then be invited to attend a measurement visit at the University of Bath for baseline assessments of fitness, blood pressure, physical activity level, and wellbeing in week 0. All participants will then enrol onto PreActiv's website, and a six-week, thrice weekly prehabilitation programme will be created for them based on their mobility and fitness level. Measurements at the University of Bath will be repeated in week 7 to assess the preliminary efficacy of PreActiv's digital prehabilitation.

Feasibility outcomes will be used to inform the design of a potential future randomised-controlled trial measuring change to cardiorespiratory fitness as the primary outcome. The decision to progress to a randomised-controlled trial will be based on pre-defined progression criteria for adherence and retention in this pilot study. In addition, participant feedback will be used to refine the study design and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Planned for major elective surgery ≥10 weeks from time of recruitment Major or complex surgery examples in NICE guideline NG45 'Routine preoperative tests for elective surgery' provides appropriate examples that are relevant to the patient cohort at the Royal United Hospitals Bath NHS Foundation Trust (RUH). We have extrapolated from these examples a list of surgical procedures that qualify as major or complex surgery and are carried out at the RUH. This list is not exhaustive but provides a range of procedures that are applicable for example: laparotomy, joint replacement, total abdominal hysterectomy, nephrectomy, neck dissection, parotidectomy, endoscopic resection of prostate, thyroidectomy.
* Aged ≥50 years

Exclusion Criteria:

* Surgery scheduled in <10 weeks
* Any relative or absolute contraindications to undertake an exercise test as described by the American College of Sports Medicine (ACSM, 2022) and the American Heart Association (Fletcher et al., 2013)
* Unsuitable to increase physical activity level as determined by Physical Activity Readiness Questionnaire (PAR-Q)
* Uncontrolled or poorly-controlled lung condition, diabetes, or seizures
* Recent (<12 months) cardiovascular events needing hospital admission
* Ongoing infection or wound making this programme hazardous for the patient
* Unable to access technology required to use the PreActiv digital platform
* Currently meeting World Health Organisation (WHO) physical activity guidelines of 75- 300 minutes of moderate to vigorous intensity physical activity per week, plus twice-weekly muscle strengthening activities
* Unable to understand explanations and/or provide informed consent
* Unable to understand written or spoken English, and without ongoing access to an interpreter
* Any condition and/or behaviour that would pose undue personal risk or introduce bias into the study
* Currently enrolled in another research trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alec Snow, MBChB, Principal Investigator — Royal United Hospitals Bath NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath, Somerset
  - University of Bath, Bath, Somerset

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed between 19th February 2024 and 19th June 2024. Recruitment took place within the preoperative assessment clinic at the Royal United Hospitals Bath NHS Foundation Trust.
Period: Baseline measurements
Arm/Group | Six weeks of digital prehabilitation
Started | 35
Completed | 31
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Expedited surgery | 1
Period: Intervention period
Arm/Group | Six weeks of digital prehabilitation
Started | 31
Commenced intervention | 28
Completed | 24
Not Completed | 7
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Expedited surgery | 1
Not completed — Adverse Event | 1
Period: Follow-up measurements
Arm/Group | Six weeks of digital prehabilitation
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Six Weeks of Digital Prehabilitation
Number analyzed (Participants) | 24
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 69 [65 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 24
Surgery type [Count of Participants; unit: Participants]
  Knee replacement | 3
  Hip replacement | 3
  Parathyroidectomy | 3
  Hernia repair | 3
  Thyroidectomy | 2
  Vaginal prolapse repair | 2
  Hysterectomy | 2
  Knee revision | 1
  Hip revision | 1
  Cholecystectomy | 1
  Prostatectomy | 1
  Ovarian cystectomy | 1
  Ureteral reimplantation | 1
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 29.1 [23.9 to 31.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited
Description: The number of patients invited that provide written informed consent, with percentage calculated
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 65
Participants | 35

2. Primary Outcome: Number of Participants Interested in Participating
Description: The number of patients invited that are willing to be screened for eligibility, with percentage calculated
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 65
Participants | 39

3. Primary Outcome: Number of Participants That Passed Screening
Description: The number of willing patients that pass screening for eligibility, with percentage calculated
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 39
Participants | 35

4. Primary Outcome: Number of Adherent Participants
Description: The number of participants who complete all exercise sessions, with percentage calculated
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
Participants | 21

5. Secondary Outcome: Cardiorespiratory Fitness
Description: Assessed via a maximal cardiopulmonary exercise test performed on a cycle ergometer, with measurements of VO2peak (ml/kg/min) and ventilatory threshold (ml/kg/min) derived.
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Population: 21/24 participants completed cardiopulmonary exercise testing.
Measure: Median (Inter-Quartile Range); unit: ml/kg/min
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 21
ml/kg/min
  Peak oxygen uptake (pre-post change) | 0.3 [-0.7 to 1.2]
  Ventilatory threshold (pre-post change) | 0.0 [-1.0 to 2.5]

6. Secondary Outcome: Resting Blood Pressure
Description: Three measurements were made after 15 minutes seated rest using an automated sphygmomanometer, with the average (mean) of the three measurements reported (mmHg)
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
mmHg
  Systolic blood pressure (pre-post change) | 1 [-10 to 12]
  Diastolic blood pressure (pre-post change) | 1 [-3 to 5]

7. Secondary Outcome: Resting Heart Rate
Description: Three measurements were made after 15 minutes seated rest using an automated sphygmomanometer, with the average (mean) of the three measurements reported (bpm)
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Measure: Median (Inter-Quartile Range); unit: beats/minute
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
beats/minute | -2 [-7 to 4]

8. Secondary Outcome: Physical Activity Level
Description: Assessed via International Physical Activity Questionnaire (IPAQ) short-form. After data processing, the highest possible score is 25,704 MET-minutes/week and the lowest possible score is 0 MET-minutes/week. A higher score is favourable as it indicates a higher physical activity level.
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Population: 20/24 participants provided complete IPAQ-short form responses for calculation of total physical activity.
Measure: Median (Inter-Quartile Range); unit: MET-minutes/week
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 20
MET-minutes/week | 852 [-53 to 2292]

9. Secondary Outcome: Anxiety and Depression
Description: Assessed via Hospital Anxiety and Depression Scale (HADS). The highest possible score is 21 and the lowest possible score is 0 for both the anxiety and depression sub-scores. A lower score is favourable as it indicates lower anxiety/depression.
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Measure: Median (Inter-Quartile Range); unit: Points
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
Points
  Anxiety (pre-post change) | -1 [-2 to 0]
  Depression (pre-post change) | -1 [-1 to 0]

10. Secondary Outcome: Quality of Life EQ-5D Visual Analogue Scale
Description: Assessed via EuroQol EQ-5D visual analogue scale, with a highest possible score of 100 and a lowest possible score of 0. A higher score is favourable as it indicates better quality of life.
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7)
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
Percentage | 5 [0 to 15]

11. Secondary Outcome: 1-minute Sit-to-stand Test
Description: Assessed via the number of repetitions completed during a 1-minute sit-to-stand test.
Time Frame: Change from pre-intervention (week 0) to post-intervention (week 7).
Population: 19/24 participants completed 1-minute sit-to-stand testing.
Measure: Median (Inter-Quartile Range); unit: Repetitions
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 19
Repetitions | 11 [6 to 14]

12. Other Pre Specified Outcome: Carbon Emissions Avoided With Home-based vs. Face-to-face Prehabilitation
Description: An estimation of the carbon emissions avoided by performing prehabilitation at home via PreActiv's digital prehabilitation compared to the estimated hypothetical emissions associated with participants travelling to the hospital three times per week for six weeks for face-to-face prehabilitation. Publicly-available carbon emissions data will be used for calculations.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: Kilograms of carbon emissions avoided
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
Kilograms of carbon emissions avoided | 44 [13 to 63]

13. Primary Outcome: Percentage of Compliant Exercise Sessions
Description: The percentage of exercise sessions that are completed as prescribed in terms of intensity, duration, and type of exercise
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 24
Percentage | 79 [68 to 90]

14. Primary Outcome: Number of Participants Retained
Description: The number of patients that enrol into the study who complete follow-up measurements, with percentage calculated
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Six weeks of digital prehabilitation
Number analyzed (Participants) | 35
Participants | 24

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, an average of 8 weeks
Arm/Group | Six weeks of digital prehabilitation
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Six weeks of digital prehabilitation (N=35)
Myocardial infarction (onset at work) (Cardiac disorders) | 1 — Assessed by the research team as not related to the intervention and reported to Sponsor. Pre-existing cardiac history. Onset of symptoms whilst at work. Successful treatment, but withdrawn from study as no longer eligible.
Diverticulitis (Gastrointestinal disorders) | 1 — Assessed by the research team as not related to the intervention and reported to Sponsor. Diverticulitis was pre-existing. Treatment in hospital only required due to presenting out-of-hours. Patient discharged the next day and completed study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Six weeks of digital prehabilitation (N=35)
Infectious illness (e.g., cold/flu) (Respiratory, thoracic and mediastinal disorders) | 2 — Exercise session delayed due to infectious illness (e.g., cold/flu).
Injury sustained at work (Musculoskeletal and connective tissue disorders) | 2 — Exercise session delayed due to injuries sustained at work.
Flare-up of fibromyalgia (Nervous system disorders) | 1 — Exercise session delayed due to flare-up of fibromyalgia symptoms.
Diverticulitis (Gastrointestinal disorders) | 1 — Exercise session delayed due to diverticulitis symptoms.

LIMITATIONS AND CAVEATS:
The lack of control group and small sample size precludes our ability to definitively attribute any effects on fitness, health, and wellbeing to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT06137781/Prot_SAP_000.pdf